CLINICAL TRIAL: NCT01012882
Title: A Multicenter Randomized DBPC Trial to Evaluate Efficacy and Safety of Sublingual Immunotherapy (SLIT) With Allergen Extracts From Pollen in Patients With Seasonal Allergic Rhinitis
Brief Title: Efficacy and Safety of Sublingual Immunotherapy (SLIT)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Roxall Medizin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLG-2009-005B
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sublingual Immunotherapy; Allergens

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- sublingual application of allergen extract (Experimental)
  Interventions: Biological: sublingual immunotherapy with allergen extract
- sublingual application of placebo (Placebo Comparator)
  Interventions: Biological: sublingual immunotherapy with placebo

INTERVENTIONS:
Biological: sublingual immunotherapy with allergen extract — sublingual application
  Arms: sublingual application of allergen extract
Biological: sublingual immunotherapy with placebo — sublingual application
  Arms: sublingual application of placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of specific sublingual immunotherapy (SLIT) with allergen extracts in patients suffering from seasonal allergic rhinitis .

ELIGIBILITY:
Inclusion Criteria:

* Positive history of allergen specific seasonal allergic rhinitis
* Positive screening skin prick test (wheal diameter > 3 mm)
* Compliance and ability of the patient to complete a Diary Card for self-evaluating of the symptoms and antisymptomatic medication
* Signed and dated patient´s Informed Consent,

Exclusion Criteria:

* Previous immunotherapy within the last 3 years,
* Simultaneous participation in other clinical trials,
* Other reasons contra-indicating an inclusion into the trial according to the investigator´s estimation (e.g. poor compliance),
* Auto-immune disorders,
* Severe chronic inflammatory diseases,
* Malignancy,
* Alcohol abuse,
* Existing or intended pregnancy, lactation and/or lack of adequate contraceptive protection,
* Treatment with beta-blockers (incl. local application) and/or other contra-indicated drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Symptom and medication score | 1 year

SECONDARY OUTCOMES:
Safety of the treatment | 1 year
Documentation of adverse events | 1 year
Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | 1 year
Clinical global improvement | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Roxall Medizin, Hamburg, Germany